CLINICAL TRIAL: NCT06791850
Title: Sustaining Home Palliative Care for Patients With Heart Failure (HF) and Their Family Caregivers in Rural Appalachia: A Mixed Methods Randomized Clinical Trial (RCT).
Brief Title: Sustaining Home Heart Failure Palliative Care in Rural Appalachia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: West Virginia University (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Ubolrat Piamjariyakul, Associate Dean for Research and Scholarship, West Virginia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2408021376; R01NR021630 (NIH)
Record Dates: First submitted 2025-01-19; First posted 2025-01-24 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-04

CONDITIONS: Heart Failure NYHA Class III; Heart Failure NYHA Class IV
Keywords: advanced heart failure; home palliative care; family caregiver; rural Appalachia

STUDY DESIGN:
Intervention Model Description: This study is a low-risk randomized control trial design to test the outcomes of the HF-FamPALhomeCARE bundled intervention with advanced HF patients and their primary family caregivers in the control group.
Who Masked: Care Provider, Outcomes Assessor
Masking Description: Care provider and outcome assessor including data collectors will be blinded to group assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Participants in control group receive standard care which is routine HF instruction at primary providers or specialist's clinic appointments.
- HF-FamPALhomeCARE (Experimental): HF-FamPALcare intervention group will receive standard care plus 2 home visits and 3 bi-weekly telephone calls on HF home EOLPC care, and follow-up telephone calls at 3, 6, 9, and 12 months.
  Interventions: Behavioral: HF-FamPALhomeCARE

INTERVENTIONS:
Behavioral: HF-FamPALhomeCARE — Participants in HF-FamPALhomeCARE Intervention group receive standard care plus 2 home visits, 3 bi-weekly telephone call on HF home EOLPC care, and follow-up telephone calls at 3, 6, 9, and 12 months.
  Arms: HF-FamPALhomeCARE

SUMMARY:
The aim of this mixed methods randomized controlled trial is to test the integrated nurse-led intervention bundle for family home care management of end-stage heart failure and palliative care in rural Appalachia. This intervention bundle is designed to address rural disparities in access to health care, with the help of the faith-based nurses and local volunteer visiting neighbors.

DETAILED DESCRIPTION:
This study uses a randomized control trial (RCT) design to test the integrated nurse-led intervention bundle of home palliative care intervention (HF-FamPALhomeCARE) for patients with heart failure (HF) and their family caregivers. (104 patient-family caregiver dyads).

The researcher will compare HF-FamPALhomeCARE to the standard control group to see if the participants in HF-FamPALhomeCARE group will report better health outcomes than the standard control group at the completion of the study at 12 months.

Aim 1: Compared to the control group at 3, 6, 9 months, and 1-year follow-up:

Hypothesis 1a. The patients in the intervention group will have higher scores on HF-related health quality-of-life measure and on the World Health Organization (WHO) aging functional health well-being scale.

Hypothesis 1b. The family caregivers in the intervention group will have higher scores on the World Health Organization (WHO) aging functional health well-being scale.

Aim 2: Compared to the control group at 3, 6, 9 months, and 1-year follow-up:

Hypothesis 2a. The patients in the intervention group will have (a) lower depression and anxiety scores and (b) higher numbers of signed EOL advance directives.

Hypothesis 2b. The family caregivers in the intervention group will have (a) lower depression and anxiety scores, (b) lower home caregiving burden scores, and (c) improved home HF EOLPC preparedness and improved home palliative care scores.

All participants receive standard care, which is routine HF instruction from their care providers. The HF-FamPALhomeCARE group receives 5-session intervention includes 2 home visits, and 3 bi-weekly telephone calls on HF home EOLPC care. Three follow-up telephone calls will be provided at 3, 6, 9, and 12 months. Control subjects will receive the same HF home care information after 12-month. Data collection for both groups are conducted at baseline, 3, 6, 9, and 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients' age between 50 to 80 years with advanced HF (NYHA III or IV), diagnosed by physician
2. Caregivers' age between 45 to 80 years.
3. Alert and consent to participate
4. Able to read and understand English

Exclusion Criteria:

1. Already received or are on a waiting list for a heart transplant or left ventricular assist device (LVAD)
2. Diagnosed with a terminal illness or dementia, such as Alzheimer's disease

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2028-04 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Patient's Kansas City Cardiomyopathy Questionnaire (KCCQ-12) | Baseline
  Measures patients' Heart Failure (HF) status & physical function status. Each item is scored on a scale from 0 to 4 or 0 to 5, depending on the question. The overall score range is 0-100 with a higher score indicating better HF health status.
Patient's Kansas City Cardiomyopathy Questionnaire (KCCQ-12) | 3 Month Follow up
  Measures patients' Heart Failure (HF) status & physical function status. Each item is scored on a scale from 0 to 4 or 0 to 5, depending on the question. The overall score range is 0-100 with a higher score indicating better HF health status.
Patient's Kansas City Cardiomyopathy Questionnaire (KCCQ-12) | 6 Month Follow up
  Measures patients' Heart Failure (HF) status & physical function status. Each item is scored on a scale from 0 to 4 or 0 to 5, depending on the question. The overall score range is 0-100 with a higher score indicating better HF health status.
Patient's Kansas City Cardiomyopathy Questionnaire (KCCQ-12) | 9 Month Follow up
  Measures patients' Heart Failure (HF) status & physical function status. Each item is scored on a scale from 0 to 4 or 0 to 5, depending on the question. The overall score range is 0-100 with a higher score indicating better HF health status.
Patient's Kansas City Cardiomyopathy Questionnaire (KCCQ-12) | 12 Month Follow Up
  Measures patients' Heart Failure (HF) status & physical function status. Each item is scored on a scale from 0 to 4 or 0 to 5, depending on the question. The overall score range is 0-100 with a higher score indicating better HF health status.
Patient--World Health Organization Quality of life Questionnaire | Baseline
  Self-assessment that measures patient's function health and well-being. Score range is 0-100 with a higher score indicating better health function and well-being.
Patient--World Health Organization Quality of life Questionnaire | 3 Month Follow up
  Self-assessment that measures patient's function health and well-being. Score range is 0-100 with a higher score indicating better health function and well-being.
Patient--World Health Organization Quality of life Questionnaire | 6 Month Follow up
  Self-assessment that measures patient's function health and well-being. Score range is 0-100 with a higher score indicating better health function and well-being.
Patient--World Health Organization Quality of life Questionnaire | 9 Month Follow up
  Self-assessment that measures patient's function health and well-being. Score range is 0-100 with a higher score indicating better health function and well-being.
Patient--World Health Organization Quality of life Questionnaire | 12 Month Follow up
  Self-assessment that measures patient's function health and well-being. Score range is 0-100 with a higher score indicating better health function and well-being.
Caregiver--World Health Organization Quality of life Questionnaire | Baseline
  Self-assessment that measures patient's function health and well-being. Score range is 0-100 with a higher score indicating better health function and well-being.
Caregiver--World Health Organization Quality of life Questionnaire | 3 Month Follow up
  Self-assessment that measures patient's function health and well-being. Score range is 0-100 with a higher score indicating better health function and well-being.
Caregiver--World Health Organization Quality of life Questionnaire | 6 Month Follow up
  Self-assessment that measures patient's function health and well-being. Score range is 0-100 with a higher score indicating better health function and well-being.
Caregiver--World Health Organization Quality of life Questionnaire | 9 Month Follow up
  Self-assessment that measures patient's function health and well-being. Score range is 0-100 with a higher score indicating better health function and well-being.
Caregiver--World Health Organization Quality of life Questionnaire | 12 Month Follow up
  Self-assessment that measures patient's function health and well-being. Score range is 0-100 with a higher score indicating better health function and well-being.

SECONDARY OUTCOMES:
Patient--Patient Health Questionnaire-9 (PHQ-9) | Baseline
  Patient Assessed: The Patient Health Questionnaire-9 (PHQ-9) is a self-administered tool used to screen, diagnose, and measure the severity of depression. It consists of nine questions with each question scored from 0 to 3 (0: Not at all, 1: Several days, 2: More than half the days, 3: Nearly every day). The total score ranges from 0 to 27, with higher scores indicating greater depressive symptoms.
Patient--Patient Health Questionnaire-9 (PHQ-9) | 3 Month Follow up
  Patient Assessed: The Patient Health Questionnaire-9 (PHQ-9) is a self-administered tool used to screen, diagnose, and measure the severity of depression. It consists of nine questions with each question scored from 0 to 3 (0: Not at all, 1: Several days, 2: More than half the days, 3: Nearly every day). The total score ranges from 0 to 27, with higher scores indicating greater depressive symptoms.
Patient--Patient Health Questionnaire-9 (PHQ-9) | 6 Month Follow up
  Patient Assessed: The Patient Health Questionnaire-9 (PHQ-9) is a self-administered tool used to screen, diagnose, and measure the severity of depression. It consists of nine questions with each question scored from 0 to 3 (0: Not at all, 1: Several days, 2: More than half the days, 3: Nearly every day). The total score ranges from 0 to 27, with higher scores indicating greater depressive symptoms.
Patient--Patient Health Questionnaire-9 (PHQ-9) | 9 Month Follow up
  Patient Assessed: The Patient Health Questionnaire-9 (PHQ-9) is a self-administered tool used to screen, diagnose, and measure the severity of depression. It consists of nine questions with each question scored from 0 to 3 (0: Not at all, 1: Several days, 2: More than half the days, 3: Nearly every day). The total score ranges from 0 to 27, with higher scores indicating greater depressive symptoms.
Patient--Patient Health Questionnaire-9 (PHQ-9) | 12 Month Follow up
  Patient Assessed: The Patient Health Questionnaire-9 (PHQ-9) is a self-administered tool used to screen, diagnose, and measure the severity of depression. It consists of nine questions with each question scored from 0 to 3 (0: Not at all, 1: Several days, 2: More than half the days, 3: Nearly every day). The total score ranges from 0 to 27, with higher scores indicating greater depressive symptoms.
Caregiver--Patient Health Questionnaire-9 (PHQ-9) | Baseline
  Caregiver Assessed: The Patient Health Questionnaire-9 (PHQ-9) is a self-administered tool used to screen, diagnose, and measure the severity of depression. It consists of nine questions with each question scored from 0 to 3 (0: Not at all, 1: Several days, 2: More than half the days, 3: Nearly every day). The total score ranges from 0 to 27, with higher scores indicating greater depressive symptoms.
Caregiver--Patient Health Questionnaire-9 (PHQ-9) | 3 Month Follow up
  Caregiver Assessed: The Patient Health Questionnaire-9 (PHQ-9) is a self-administered tool used to screen, diagnose, and measure the severity of depression. It consists of nine questions with each question scored from 0 to 3 (0: Not at all, 1: Several days, 2: More than half the days, 3: Nearly every day). The total score ranges from 0 to 27, with higher scores indicating greater depressive symptoms.
Caregiver--Patient Health Questionnaire-9 (PHQ-9) | 6 Month Follow up
  Caregiver Assessed: The Patient Health Questionnaire-9 (PHQ-9) is a self-administered tool used to screen, diagnose, and measure the severity of depression. It consists of nine questions with each question scored from 0 to 3 (0: Not at all, 1: Several days, 2: More than half the days, 3: Nearly every day). The total score ranges from 0 to 27, with higher scores indicating greater depressive symptoms.
Caregiver--Patient Health Questionnaire-9 (PHQ-9) | 9 Month Follow up
  Caregiver Assessed: The Patient Health Questionnaire-9 (PHQ-9) is a self-administered tool used to screen, diagnose, and measure the severity of depression. It consists of nine questions with each question scored from 0 to 3 (0: Not at all, 1: Several days, 2: More than half the days, 3: Nearly every day). The total score ranges from 0 to 27, with higher scores indicating greater depressive symptoms.
Caregiver--Patient Health Questionnaire-9 (PHQ-9) | 12 Month Follow up
  Caregiver Assessed: The Patient Health Questionnaire-9 (PHQ-9) is a self-administered tool used to screen, diagnose, and measure the severity of depression. It consists of nine questions with each question scored from 0 to 3 (0: Not at all, 1: Several days, 2: More than half the days, 3: Nearly every day). The total score ranges from 0 to 27, with higher scores indicating greater depressive symptoms.
Patient--Generalized anxiety disorder (GAD-7) | Baseline
  Patient Assessed: The Generalized Anxiety Disorder 7-item (GAD-7) scale is a self-administered questionnaire designed to screen for and measure the severity of generalized anxiety disorder (GAD). It consists of seven items that assess how often the respondent has been bothered by various anxiety symptoms. Each item is scored on a scale from 0 to 3 (0: Not at all, 1: Several days, 2: More than half the days, 3: Nearly every day). Overall score range of 0-21 with a higher score indicating greater anxiety symptoms.
Patient--Generalized anxiety disorder (GAD-7) | 3 Month Follow up
  Patient Assessed: The Generalized Anxiety Disorder 7-item (GAD-7) scale is a self-administered questionnaire designed to screen for and measure the severity of generalized anxiety disorder (GAD). It consists of seven items that assess how often the respondent has been bothered by various anxiety symptoms. Each item is scored on a scale from 0 to 3 (0: Not at all, 1: Several days, 2: More than half the days, 3: Nearly every day). Overall score range of 0-21 with a higher score indicating greater anxiety symptoms.
Patient--Generalized anxiety disorder (GAD-7) | 6 Month Follow up
  Patient Assessed: The Generalized Anxiety Disorder 7-item (GAD-7) scale is a self-administered questionnaire designed to screen for and measure the severity of generalized anxiety disorder (GAD). It consists of seven items that assess how often the respondent has been bothered by various anxiety symptoms. Each item is scored on a scale from 0 to 3 (0: Not at all, 1: Several days, 2: More than half the days, 3: Nearly every day). Overall score range of 0-21 with a higher score indicating greater anxiety symptoms.
Patient--Generalized anxiety disorder (GAD-7) | 9 Month Follow up
  Patient Assessed: The Generalized Anxiety Disorder 7-item (GAD-7) scale is a self-administered questionnaire designed to screen for and measure the severity of generalized anxiety disorder (GAD). It consists of seven items that assess how often the respondent has been bothered by various anxiety symptoms. Each item is scored on a scale from 0 to 3 (0: Not at all, 1: Several days, 2: More than half the days, 3: Nearly every day). Overall score range of 0-21 with a higher score indicating greater anxiety symptoms.
Patient--Generalized anxiety disorder (GAD-7) | 12 Month Follow up
  Patient Assessed: The Generalized Anxiety Disorder 7-item (GAD-7) scale is a self-administered questionnaire designed to screen for and measure the severity of generalized anxiety disorder (GAD). It consists of seven items that assess how often the respondent has been bothered by various anxiety symptoms. Each item is scored on a scale from 0 to 3 (0: Not at all, 1: Several days, 2: More than half the days, 3: Nearly every day). Overall score range of 0-21 with a higher score indicating greater anxiety symptoms.
Caregiver--Generalized anxiety disorder (GAD-7) | Baseline
  Caregiver Assessed: The Generalized Anxiety Disorder 7-item (GAD-7) scale is a self-administered questionnaire designed to screen for and measure the severity of generalized anxiety disorder (GAD). It consists of seven items that assess how often the respondent has been bothered by various anxiety symptoms. Each item is scored on a scale from 0 to 3 (0: Not at all, 1: Several days, 2: More than half the days, 3: Nearly every day). Overall score range of 0-21 with a higher score indicating greater anxiety symptoms.
Caregiver--Generalized anxiety disorder (GAD-7) | 3 Month Follow up
  Caregiver Assessed: The Generalized Anxiety Disorder 7-item (GAD-7) scale is a self-administered questionnaire designed to screen for and measure the severity of generalized anxiety disorder (GAD). It consists of seven items that assess how often the respondent has been bothered by various anxiety symptoms. Each item is scored on a scale from 0 to 3 (0: Not at all, 1: Several days, 2: More than half the days, 3: Nearly every day). Overall score range of 0-21 with a higher score indicating greater anxiety symptoms.
Caregiver--Generalized anxiety disorder (GAD-7) | 6 Month Follow up
  Caregiver Assessed: The Generalized Anxiety Disorder 7-item (GAD-7) scale is a self-administered questionnaire designed to screen for and measure the severity of generalized anxiety disorder (GAD). It consists of seven items that assess how often the respondent has been bothered by various anxiety symptoms. Each item is scored on a scale from 0 to 3 (0: Not at all, 1: Several days, 2: More than half the days, 3: Nearly every day). Overall score range of 0-21 with a higher score indicating greater anxiety symptoms.
Caregiver--Generalized anxiety disorder (GAD-7) | 9 Month Follow up
  Caregiver Assessed: The Generalized Anxiety Disorder 7-item (GAD-7) scale is a self-administered questionnaire designed to screen for and measure the severity of generalized anxiety disorder (GAD). It consists of seven items that assess how often the respondent has been bothered by various anxiety symptoms. Each item is scored on a scale from 0 to 3 (0: Not at all, 1: Several days, 2: More than half the days, 3: Nearly every day). Overall score range of 0-21 with a higher score indicating greater anxiety symptoms.
Caregiver--Generalized anxiety disorder (GAD-7) | 12 Month Follow up
  Caregiver Assessed: The Generalized Anxiety Disorder 7-item (GAD-7) scale is a self-administered questionnaire designed to screen for and measure the severity of generalized anxiety disorder (GAD). It consists of seven items that assess how often the respondent has been bothered by various anxiety symptoms. Each item is scored on a scale from 0 to 3 (0: Not at all, 1: Several days, 2: More than half the days, 3: Nearly every day). Overall score range of 0-21 with a higher score indicating greater anxiety symptoms.
Patient--Integrated Palliative care Outcome Scale (IPOS) | Baseline
  Patient reported: Integrated Palliative care Outcome Scale (IPOS) is a holistic assessment used to measure the symptoms and concerns of patients receiving palliative care. Each item is scored based on the patient's response, typically on a scale from 0 to 4 with an overall score range of 0 to 68. A higher overall score indicates more palliative care problems or concerns.
Patient--Integrated Palliative care Outcome Scale (IPOS) | 3 Month Follow up
  Patient reported: Integrated Palliative care Outcome Scale (IPOS) is a holistic assessment used to measure the symptoms and concerns of patients receiving palliative care. Each item is scored based on the patient's response, typically on a scale from 0 to 4 with an overall score range of 0 to 68. A higher overall score indicates more palliative care problems or concerns.
Patient--Integrated Palliative care Outcome Scale (IPOS) | 6 Month Follow up
  Patient reported: Integrated Palliative care Outcome Scale (IPOS) is a holistic assessment used to measure the symptoms and concerns of patients receiving palliative care. Each item is scored based on the patient's response, typically on a scale from 0 to 4 with an overall score range of 0 to 68. A higher overall score indicates more palliative care problems or concerns.
Patient--Integrated Palliative care Outcome Scale (IPOS) | 9 Month Follow up
  Patient reported: Integrated Palliative care Outcome Scale (IPOS) is a holistic assessment used to measure the symptoms and concerns of patients receiving palliative care. Each item is scored based on the patient's response, typically on a scale from 0 to 4 with an overall score range of 0 to 68. A higher overall score indicates more palliative care problems or concerns.
Patient--Integrated Palliative care Outcome Scale (IPOS) | 12 Month Follow up
  Patient reported: Integrated Palliative care Outcome Scale (IPOS) is a holistic assessment used to measure the symptoms and concerns of patients receiving palliative care. Each item is scored based on the patient's response, typically on a scale from 0 to 4 with an overall score range of 0 to 68. A higher overall score indicates more palliative care problems or concerns.
Caregiver--Integrated Palliative care Outcome Scale (IPOS) | Baseline
  Caregiver reported: Integrated Palliative care Outcome Scale (IPOS) is a holistic assessment used to measure the symptoms and concerns of caregivers receiving palliative care. Each item is scored based on the patient's response, typically on a scale from 0 to 4 with an overall score range of 0 to 68. A higher overall score indicates more palliative care problems or concerns.
Caregiver--Integrated Palliative care Outcome Scale (IPOS) | 3 Month Follow up
  Caregiver reported: Integrated Palliative care Outcome Scale (IPOS) is a holistic assessment used to measure the symptoms and concerns of caregivers receiving palliative care. Each item is scored based on the patient's response, typically on a scale from 0 to 4 with an overall score range of 0 to 68. A higher overall score indicates more palliative care problems or concerns.
Caregiver--Integrated Palliative care Outcome Scale (IPOS) | 6 Month Follow up
  Caregiver reported: Integrated Palliative care Outcome Scale (IPOS) is a holistic assessment used to measure the symptoms and concerns of caregivers receiving palliative care. Each item is scored based on the patient's response, typically on a scale from 0 to 4 with an overall score range of 0 to 68. A higher overall score indicates more palliative care problems or concerns.
Caregiver--Integrated Palliative care Outcome Scale (IPOS) | 9 Month Follow up
  Caregiver reported: Integrated Palliative care Outcome Scale (IPOS) is a holistic assessment used to measure the symptoms and concerns of caregivers receiving palliative care. Each item is scored based on the patient's response, typically on a scale from 0 to 4 with an overall score range of 0 to 68. A higher overall score indicates more palliative care problems or concerns.
Caregiver--Integrated Palliative care Outcome Scale (IPOS) | 12 Month Follow up
  Caregiver reported: Integrated Palliative care Outcome Scale (IPOS) is a holistic assessment used to measure the symptoms and concerns of caregivers receiving palliative care. Each item is scored based on the patient's response, typically on a scale from 0 to 4 with an overall score range of 0 to 68. A higher overall score indicates more palliative care problems or concerns.
Patient--Functional Assessment of Chronic Illness Therapy - Spiritual Well-Being 12 Item Scale (FACIT-12) | Baseline
  Assessment of spiritual well-being of patient managing chronic health conditions. Consists of 12 items with each item rated on a 5-point Likert scale, ranging from 0 (not at all) to 4 (very much). Total score range is 0 to 48 with higher score indicating higher spiritual well-being.
Patient--Functional Assessment of Chronic Illness Therapy - Spiritual Well-Being 12 Item Scale (FACIT-12) | 3 Month Follow up
  Assessment of spiritual well-being of patient managing chronic health conditions. Consists of 12 items with each item rated on a 5-point Likert scale, ranging from 0 (not at all) to 4 (very much). Total score range is 0 to 48 with higher score indicating higher spiritual well-being.
Patient--Functional Assessment of Chronic Illness Therapy - Spiritual Well-Being 12 Item Scale (FACIT-12) | 6 Month Follow up
  Assessment of spiritual well-being of patient managing chronic health conditions. Consists of 12 items with each item rated on a 5-point Likert scale, ranging from 0 (not at all) to 4 (very much). Total score range is 0 to 48 with higher score indicating higher spiritual well-being.
Patient--Functional Assessment of Chronic Illness Therapy - Spiritual Well-Being 12 Item Scale (FACIT-12) | 9 Month Follow up
  Assessment of spiritual well-being of patient managing chronic health conditions. Consists of 12 items with each item rated on a 5-point Likert scale, ranging from 0 (not at all) to 4 (very much). Total score range is 0 to 48 with higher score indicating higher spiritual well-being.
Patient--Functional Assessment of Chronic Illness Therapy - Spiritual Well-Being 12 Item Scale (FACIT-12) | 12 Month Follow up
  Assessment of spiritual well-being of patient managing chronic health conditions. Consists of 12 items with each item rated on a 5-point Likert scale, ranging from 0 (not at all) to 4 (very much). Total score range is 0 to 48 with higher score indicating higher spiritual well-being.
Caregiver--Functional Assessment of Chronic Illness Therapy - Spiritual Well-Being 12 Item Scale (FACIT-12) | Baseline
  Assessment of spiritual well-being of caregiver managing chronic health conditions. Consists of 12 items with each item rated on a 5-point Likert scale, ranging from 0 (not at all) to 4 (very much). Total score range is 0 to 48 with higher score indicating higher spiritual well-being.
Caregiver--Functional Assessment of Chronic Illness Therapy - Spiritual Well-Being 12 Item Scale (FACIT-12) | 3 Month Follow up
  Assessment of spiritual well-being of caregiver managing chronic health conditions. Consists of 12 items with each item rated on a 5-point Likert scale, ranging from 0 (not at all) to 4 (very much). Total score range is 0 to 48 with higher score indicating higher spiritual well-being.
Caregiver--Functional Assessment of Chronic Illness Therapy - Spiritual Well-Being 12 Item Scale (FACIT-12) | 6 Month Follow up
  Assessment of spiritual well-being of caregiver managing chronic health conditions. Consists of 12 items with each item rated on a 5-point Likert scale, ranging from 0 (not at all) to 4 (very much). Total score range is 0 to 48 with higher score indicating higher spiritual well-being.
Caregiver--Functional Assessment of Chronic Illness Therapy - Spiritual Well-Being 12 Item Scale (FACIT-12) | 9 Month Follow up
  Assessment of spiritual well-being of caregiver managing chronic health conditions. Consists of 12 items with each item rated on a 5-point Likert scale, ranging from 0 (not at all) to 4 (very much). Total score range is 0 to 48 with higher score indicating higher spiritual well-being.
Caregiver--Functional Assessment of Chronic Illness Therapy - Spiritual Well-Being 12 Item Scale (FACIT-12) | 12 Month Follow up
  Assessment of spiritual well-being of caregiver managing chronic health conditions. Consists of 12 items with each item rated on a 5-point Likert scale, ranging from 0 (not at all) to 4 (very much). Total score range is 0 to 48 with higher score indicating higher spiritual well-being.
The Zarit Burden Interview (ZBI-12) | Baseline
  The ZBI-12 consists of 12 questions that caregivers answer based on how often they experience certain feelings related to their caregiving role. Each question is scored on a scale from 0 (never) to 4 (nearly always), with the total score ranging from 0 to 48 with a higher score indicating greater burden.
The Zarit Burden Interview (ZBI-12) | 3 Month Follow up
  The ZBI-12 consists of 12 questions that caregivers answer based on how often they experience certain feelings related to their caregiving role. Each question is scored on a scale from 0 (never) to 4 (nearly always), with the total score ranging from 0 to 48 with a higher score indicating greater burden.
The Zarit Burden Interview (ZBI-12) | 6 Month Follow up
  The ZBI-12 consists of 12 questions that caregivers answer based on how often they experience certain feelings related to their caregiving role. Each question is scored on a scale from 0 (never) to 4 (nearly always), with the total score ranging from 0 to 48 with a higher score indicating greater burden.
The Zarit Burden Interview (ZBI-12) | 9 Month Follow up
  The ZBI-12 consists of 12 questions that caregivers answer based on how often they experience certain feelings related to their caregiving role. Each question is scored on a scale from 0 (never) to 4 (nearly always), with the total score ranging from 0 to 48 with a higher score indicating greater burden.
The Zarit Burden Interview (ZBI-12) | 12 Month Follow up
  The ZBI-12 consists of 12 questions that caregivers answer based on how often they experience certain feelings related to their caregiving role. Each question is scored on a scale from 0 (never) to 4 (nearly always), with the total score ranging from 0 to 48 with a higher score indicating greater burden.

CONTACTS AND LOCATIONS:
Overall Officials: Ubolrat Piamjariyakul, Principal Investigator — West Virginia University School of Nursing
Locations (1):
- West Virginia University Hospital, Morgantown, West Virginia, United States

IPD SHARING:
Plan to Share IPD: Yes
To enhance the transparency, and reproducibility of the research, the de-identified dataset, project data descriptions, and statistical models generated by this R01 will be shared. These data will be shared in the appropriate NIH repository the National Archive of Computerized Data on Aging (NACDA) hosted by ICPSR. The description of the data management plan is also submitted.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Study protocol and SAP will be shared via ClinicalTrials.gov and published protocol manuscript.
  The Analysis codes will be made available at the end of the project period and at the time of publication.
Access Criteria: There is no public access to the database during the trial period. This project's scientific data will be available on the NACDA NIH Repository 5 years after the end of the funding period.

REFERENCES:
- [Derived] Piamjariyakul U, Young S, Smothers A, Wen S, Navia RO, Sokos G, Hendrickson AE, Fink P, Niland D, Hottle M, Giolzetti AC, Smith CE. Study protocol of sustaining home palliative care for patients with Heart Failure (HF) and their family caregivers in rural Appalachia: a mixed methods randomized clinical trial. BMC Palliat Care. 2025 Mar 7;24(1):56. doi: 10.1186/s12904-025-01680-y. PMID 40055735